CLINICAL TRIAL: NCT05539690
Title: Effect of Balance Training on White Matter Tracts in Healthy Elderly Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Youngkook Kim, Assistant professor, The Catholic University of Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SC22FISI0069
Record Dates: First submitted 2022-09-11; First posted 2022-09-14 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Postural Balance; Neuronal Plasticity; Elderly Population
Keywords: Postural Balance; White Matter; Neuronal Plasticity; Elderly Population; Rehabilitation; Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balance training group (Experimental): A single training group
  Interventions: Behavioral: Balance training

INTERVENTIONS:
Behavioral: Balance training — * Step-by-step training (5 levels)
  * 30 minute per training
  * 3 times per week
  * 4 weeks

SUMMARY:
Balance impairment increases the risk of falling and is associated with a fear of falling and immobility. Balance impairment can ultimately affect the morbidity of cardiovascular disease, cognitive impairment, and mortality, especially in an older population. Among the multiple types of exercise, balance training is the most effective in preventing falls. This study aims to investigate white matter plasticity in healthy elderly population, based on stepwise balance training. Healthy elderly participants will undergo four weeks of balance training. The investigators will analyze longitudinal changes in the microstructural integrity of the white matter tracts pre- and post-training.

DETAILED DESCRIPTION:
Balance is an essential element of daily living. Balance impairment increases the risk of falling and is associated with a fear of falling and immobility. Balance impairment can ultimately affect the morbidity of cardiovascular disease, cognitive impairment, and mortality, especially in an older population. Among the multiple types of exercise, balance training is the most effective in preventing falls. Specific structures of the brain are highly associated with balance, and the integration of functions from these structures maintains balance function.

Training-induced behavioral changes accompany white matter plasticity. White matter plasticity by practicing expert skills has been of particular interest because characteristic changes in white matter are expected to occur through repetitive and intensive motor skill training. Training-induced white matter plasticity regarding balance is less understood in the healthy adult population. Previous neuroimaging studies have focused on elucidating the cross-sectional associations between balance function and disease-specific characteristics in various clinical populations, such as patients with stroke, traumatic brain injury, Parkinson's disease, and other neurodegenerative diseases.

Developing neuroimaging biomarkers is essential to provide individualized training or rehabilitation intervention and to evaluate its efficacy. Diffusion tensor imaging is a sensitive neuroimaging tool to detect myelin change quantitatively in human white matter in vivo. DTI is used to measure water molecules' diffusion anisotropy, called fractional anisotropy (FA).

This study will explore white matter plasticity in a healthy elderly population which practices stepwise balance training for 4 weeks. The investigators adopt a longitudinal design to contrast the neuroplastic changes in white matter tracts linked to balance function. The investigators hypothesize that balance training would change the microstructural integrity of white matter tracts associated with balance improvement.

ELIGIBILITY:
Inclusion Criteria:

* Mini-mental state examination ≥ 26
* Independent outdoor ambulator

Exclusion Criteria:

* Men/women with any metal implants in their body
* A prior history of psychopathology or a neurological disorders
* A prior history of osteoporosis, advanced osteoarthritis (K-L grade >=3), surgical history of hip or knee arthroplasty
* If any structural abnormalities are detected on their scan

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Fractional anisotropy of the motor-related white matter tracts | 4 weeks
  Measurement of the change of DTI-derived parameter before and after balance training
  1. Tracts of interest
     * Corticospinal tract (CST)
     * Cortico-ponto-cerebellar tract (CPCT)
     * Dentato-rubro-thalamo-cortical tract (DRTCT)
     * Dorsal spinocerebellar tract (DSCT)
  2. Measurement of DTI-derived parameter
     * Fractional anisotropy (FA) values of the CST, CPCT, DRTCT, and DSCT
  3. Units and scoring of the Measurement
     * FA
       * No unit.
       * The measurement ranges from 0 to 1
       * Higher scores indicate better microstructural integrity.
Community Balance & Mobility Scale | 4 weeks
  Performance measure before and after balance training
  1. Measurement
     * 13 domain
     * Unilateral stance, Tandem walking, 180° tandem pivot, Lateral foot scooting, Hopping forward, Crouch and walk, Lateral dodging, Walking & looking, Running with controlled stop, Forward to backward walking, Walk look and carry, Descending stairs, Step-ups x 1 step
  2. Scoring of the Measurement
     * No units.
     * The measurement ranges from 0 to 96
     * Higher scores indicate better postural balance and mobility.

SECONDARY OUTCOMES:
Mean diffusivity of the motor-related white matter tracts | 4 weeks
  Measurement of the change of DTI-derived parameter before and after balance training
  1. Tracts of interest
     * CST
     * CPCT
     * DRTCT
     * DSCT
  2. Measurement of DTI-derived parameter
     * Mean Diffusivity (MD) values of the CST, CPCT, DRTCT, and DSCT
  3. Units and scoring of the Measurement
     * MD
       * mm^2/second
       * There is no limit on the range (usually ranges 0.00005 - 0.0001 mm^2/second).
       * Higher scores indicate worse microstructural integrity.
Tract volume of the motor-related white matter tracts | 4 weeks
  Measurement of the change of DTI-derived parameter before and after balance training
  1. Tracts of interest
     * CST
     * CPCT
     * DRTCT
     * DSCT
  2. Measurement of DTI-derived parameter
     * Tract volume (TV) values of the CST, CPCT, DRTCT, and DSCT
  3. Units and scoring of the Measurement
     * TV
       * mm^3
       * There is no limit on the range.
       * Higher scores indicate better microstructural integrity.

CONTACTS AND LOCATIONS:
Overall Officials: Youngkook Kim, MD, PhD, Principal Investigator — Yeouido St. Mary's Hospital, College of Medicine, The Catholic University of Korea
Locations (1):
- Yeouido St. Mary's Hospital, Seoul, Yeongdeungpo-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sherrington C, Fairhall NJ, Wallbank GK, Tiedemann A, Michaleff ZA, Howard K, Clemson L, Hopewell S, Lamb SE. Exercise for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2019 Jan 31;1(1):CD012424. doi: 10.1002/14651858.CD012424.pub2. PMID 30703272
- [Result] Surgent OJ, Dadalko OI, Pickett KA, Travers BG. Balance and the brain: A review of structural brain correlates of postural balance and balance training in humans. Gait Posture. 2019 Jun;71:245-252. doi: 10.1016/j.gaitpost.2019.05.011. Epub 2019 May 6. PMID 31082657
- [Result] Scholz J, Klein MC, Behrens TE, Johansen-Berg H. Training induces changes in white-matter architecture. Nat Neurosci. 2009 Nov;12(11):1370-1. doi: 10.1038/nn.2412. Epub 2009 Oct 11. PMID 19820707
- [Result] Kim JS, Kim SH, Lim SH, Im S, Hong BY, Oh J, Kim Y. Degeneration of the Inferior Cerebellar Peduncle After Middle Cerebral Artery Stroke: Another Perspective on Crossed Cerebellar Diaschisis. Stroke. 2019 Oct;50(10):2700-2707. doi: 10.1161/STROKEAHA.119.025723. Epub 2019 Aug 26. PMID 31446886
- [Result] Kim Y, Kim SH, Hong BY, Oh J, Chang SY. Integrity of the Inferior Cerebellar Peduncle Correlates with Ambulatory Function after Hemorrhagic Stroke. J Stroke Cerebrovasc Dis. 2021 Dec;30(12):106164. doi: 10.1016/j.jstrokecerebrovasdis.2021.106164. Epub 2021 Oct 13. PMID 34655972